CLINICAL TRIAL: NCT06849388
Title: Resilience as a Journey, Not a Destination: The Feasibility of Applying HeartMath to Stress, Emotional Vitality and Sense of Coherence Among Intensive Care Units Nurses.
Brief Title: Effect of HeartMath Intervention on Stress, Emotional Vitality and Sense of Coherence
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Damanhour University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: HeartMath
Record Dates: First submitted 2025-02-22; First posted 2025-02-27 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2025-02

CONDITIONS: Stress; Coherence Sense

STUDY DESIGN:
Intervention Model Description: intervention group will used heart math intervention control group have no intervention
Who Masked: Participant
Masking Description: the participant will be masked for the intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Heart Math group (Experimental): Nurses will be included in heart math program
  Interventions: Behavioral: Heart Math program
- Control group (No Intervention): Nurses who will receive no intervention

INTERVENTIONS:
Behavioral: Heart Math program — Heart Math program is behavior intervention through several sessions
  Arms: Heart Math group

SUMMARY:
This study aims to investigate the effect of Heart math intervention program on stress, emotional vitality and sense of coherence among intensive care units Nurses

DETAILED DESCRIPTION:
This study aims to investigate the effect of Heart math intervention program on stress, emotional vitality and sense of coherence among intensive care units Nurses.

The intervention was implemented in form of 2 sessions per week according to the following 7 sessions, each session about 45- 60 minutes.

Session (1)

Aims:

Introduce Heart Math definition of stress. Assess client's current stress level.

Handouts for patients:

Handout 1 : Stress What is stress? How stress affect health? How stressed are you? What can I do about it? Session (2) Aim: Introduce concept of heart coherence

Handouts for patients:

Handout 1: Heart Coherence How dose Heart Math work? How can I create and practice physiological coherence? The Quick Coherence Technique. Handout 2: Depletion to renewal plan. Session (3)

Aims:

Teach Heart-Focused Breathing and Quick Coherence Introduce personal practice plan to use for

Handouts for patients:

Handout 1: Heart-focused breathing. Handout 2: Quick coherence technique. Handout 3: Personal practice log. Session (4)

Aims:

Assess client's current anxiety level. Review this week's homework on Personal Practice Log. Review and practice Quick Coherence Technique. Teach Heart Lock-In Technique.

Handouts for patients:

Handout 1: Anxiety Checklist. Handout 2: Quick Coherence Technique. Handout 3: Heart Lock-In Technique. Handout 3: Personal Practice Log. Session (5)

Aims:

Review this week's homework on Personal Practice Log. Review Heart-Focused Breathing and Quick Coherence Techniques. Review and practice. Heart Lock-In Technique. Teach Freeze Frame Technique.

Handouts for patients:

Handout 1: Heart Lock-In Technique. Handout 2: Freeze Frame Technique. Session (6)

Aims:

Review this week's homework on Personal Practice Log. Review Heart Lock-In and Freeze Frame Techniques. Teach Attitude Breathing Technique.

Handouts for patients:

Handout 1: Personal Practice Log. Handout 2: Freeze Frame Technique. Handout 3: Attitude Breathing Technique. Session (7)

Aims:

Review this week's homework on Attitude Breathing Technique. Teach Coherence Communication Technique.

Handouts for patients:

Handout 1: Attitude Breathing Technique. Handout 2: Coherent Communication Technique.

ELIGIBILITY:
Inclusion Criteria:

* Nurses who work in selected intensive care units and agree to participate

Exclusion Criteria:

* Nurses who refuse to participate in this study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Resilience Scale | over two months
  The Resilience Scale consisted of 25 items and a short version contained 14 items.
  The scale is a 7-point Likert type scale from 1 (Strongly disagree) to 7 (Strongly agree) for each item. Scores on the scale range from 14 to 98. The higher score indicates the ability to respond with resilience and lower score indicates lower resilience.
Personal and Organizational Quality Assessment | over two months
  It is a valid and reliable 52-item survey tool developed by the Heart Math Institute that assesses personal health, resiliency, and workplace factors impacting an organization's quality and effectiveness. It is composed of 4 primary scales (emotional vitality, organizational stress, emotional stress, and physical stress), which are further divided into 9 subscales. These scales assess elements that either enhance or impair work performance, health, well-being, and job satisfaction.
Sense of Coherence | over two months
  The Sense of Coherence scale measure the concept of sense of coherence. The short form of the Sense of Coherence scale consists of 13 items that comprise three components: comprehensibility (to which 5 items contribute), manageability (4 items), and meaningfulness (4 items). The respondents indicate agreement or disagreement on a 7-category semantic differential scale with two anchoring responses tailored to the content of each item. Five items (1, 2, 3, 5, and 7) are reversed before summing the total score. The total score can range from 13 to 91, and a higher score indicates higher coherence .

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Nursing, Damanhūr, Damanhour
  - Damanhour university, Damanhūr

IPD SHARING:
Plan to Share IPD: Undecided